CLINICAL TRIAL: NCT00617357
Title: A Multicenter, Prospective, Observational Evaluation of Repair of Infected or Contaminated Hernias (RICH) Using LTM
Brief Title: Repair of Infected or Contaminated Hernias
Acronym: RICH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LifeCell (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LFC2007.02.01
Record Dates: First submitted 2008-01-14; First posted 2008-02-18 (Estimated); Results first posted 2015-12-01 (Estimated); Last update posted 2015-12-01 (Estimated); Status verified 2015-10

CONDITIONS: Hernia
Keywords: incisional hernia; abdominal hernia repair; Ventral incisional hernia repair
MeSH Terms: conditions — Hernia; Incisional Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Strattice Reconstructive Tissue Matrix
  Interventions: Device: LTM (Strattice Reconstructive Tissue Matrix)

INTERVENTIONS:
Device: LTM (Strattice Reconstructive Tissue Matrix) — Surgical mesh

SUMMARY:
This is a prospective, multicenter, interventional, observational, open label, single arm, longitudinal evaluation of ventral incisional hernia repair using LTM in contaminated or infected sites. Three interim analyses are planned to examine the incidence of surgical site events, postoperative resumption of activities and hernia recurrence.

ELIGIBILITY:
Inclusion Criteria:

* is an adult ≥18 years old.
* has need of open abdominal incisional repair of a contaminated or infected site
* has an estimated hernia size of >9cm2 by physical exam

Exclusion Criteria:

* has a nidus of chronic colonization
* has a systemic infection at the time of repair.
* has chronic conditions: hepatic cirrhosis (w/ or w/o ascites); renal failure w/ hemo- or peritoneal dialysis; incomplete resection of malignant disease; or defined collagen disorder.
* requires chronic immunosuppressive therapy, including steroids or cytotoxic agents.
* is bedridden or otherwise non-ambulatory.
* is ASA Class 4 or 5.
* has a BMI >40.
* has conditions that would adversely affect subject safety, as per product labeling, including sensitivities to pork or porcine products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2007-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Itani, MD, Principal Investigator — Boston VA Healthcare System
Locations (15):
- United States (15):
  - University of California-San Diego Medical Center, La Jolla, California
  - Hospital of St Rafael, New Haven, Connecticut
  - Louisiana State University Health Sciences Center, New Orleans, Louisiana
  - Tulane University Medical Center, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of Missouri-Columbia Medical Center, Columbia, Missouri
  - Washington University, St Louis, Missouri
  - North Shore University Hospital-Long Island Jewish Health System, Manhasset, New York
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Baylor College of Medicine, Houston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Utah Medical Center, Salt Lake City, Utah

REFERENCES:
- [Result] Itani KM, Rosen M, Vargo D, Awad SS, Denoto G 3rd, Butler CE; RICH Study Group. Prospective study of single-stage repair of contaminated hernias using a biologic porcine tissue matrix: the RICH Study. Surgery. 2012 Sep;152(3):498-505. doi: 10.1016/j.surg.2012.04.008. Epub 2012 Jul 3. PMID 22763262
- [Derived] Rosen MJ, Denoto G, Itani KM, Butler C, Vargo D, Smiell J, Rutan R. Evaluation of surgical outcomes of retro-rectus versus intraperitoneal reinforcement with bio-prosthetic mesh in the repair of contaminated ventral hernias. Hernia. 2013 Feb;17(1):31-5. doi: 10.1007/s10029-012-0909-2. Epub 2012 Mar 14. PMID 22415440

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 83 subjects enrolled between Sep 2007 and Aug 2008 from 12 US sites and followed for 24 months following hernia repair
Pre-assignment Details: 83 subjects were enrolled, 3 were not implanted, resulting in 80 subjects implanted with device (ITT group).
Period: Overall Study
Arm/Group | Strattice Tissue Matrix
Started | 83 (83 subjects enrolled, 80 subjects received Strattice reinforcement of hernia repair)
Completed | 67 (67 subjects completed study; 7 completed early, 60 completed 24 month visit)
Not Completed | 16
Not completed — Lost to Follow-up | 7
Not completed — Death | 5
Not completed — insurance concerns | 2
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: 83 subjects enrolled, of which 80 subjects were implanted. The ITT population is defined as subjects enrolled and implanted (n=80).
Groups:
- One Arm: Strattice Reconstructive Tissue Matrix
Arm/Group | One Arm
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 47
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 71
  Black or African American | 9
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Wound Events
Description: Wound Events are defined as those events which occurred in the area of the hernia repair and the repair site, including seroma, hematoma, dehiscence, infection, abscess, fistula, and re-herniation.
Time Frame: Postoperatively up to 24 months
Population: 80 patients were enrolled and received Strattice Reconstructive Tissue Matrix to support the repair and were included in the Intent to Treat (ITT) population.
Measure: Number; unit: participants
Arm/Group | One Arm
Number analyzed (Participants) | 80
participants | 53

2. Secondary Outcome: Activities Assessment Scale (AAS)
Description: The AAS includes 13 items covering a broad sample of sedentary, movement-related and graded-intensity physical activities. Respondents are asked to rate the degree of difficulty performing each of these activities in the previous 24 hours on a 5-point scale from "No difficulty" to "Not able to do it." The AAS has three subscales: sedentary activities (items 1-4); ambulatory activities (items 6-8); work/exercise activities (items 11-13). The AAS total and subscale scores are numerically transformed to produce a range of 0-100, with higher values indicating greater functional activity.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Strattice Reconstructive Tissue Matrix: Subjects implanted with Strattice Reconstructive Tissue Matrix in the repair of infected or contaminated hernias.
  LTM (Strattice Reconstructive Tissue Matrix): Surgical mesh
Arm/Group | Strattice Reconstructive Tissue Matrix
Number analyzed (Participants) | 79
units on a scale | 69.2 (21.45)

3. Secondary Outcome: Activities Assessment Scale (AAS)
Description: The AAS includes 13 items covering a broad sample of sedentary, movement-related and graded-intensity physical activities. Respondents are asked to rate the degree of difficulty performing each of these activities in the previous 24 hours on a 5-point scale from "No difficulty" to "Not able to do it." The AAS has three subscales: sedentary activities (items 1-4); ambulatory activities (items 6-8); work/exercise activities (items 11-13). The AAS total and subscale scores are transformed to produce a range of 0-100, with higher values indicating greater functional activity.
Time Frame: 30 Days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Strattice Reconstructive Tissue Matrix
Number analyzed (Participants) | 72
units on a scale | 70.3 (19.47)

4. Secondary Outcome: Activities Assessment Scale (AAS)
Description: as for outcome 3
Time Frame: 3 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Strattice Reconstructive Tissue Matrix
Number analyzed (Participants) | 70
units on a scale | 78.2 (16.06)

5. Secondary Outcome: Activities Assessment Scale (AAS)
Description: as for outcome 3
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Strattice Reconstructive Tissue Matrix
Number analyzed (Participants) | 73
units on a scale | 85.3 (14.17)

6. Secondary Outcome: Activities Assessment Scale (AAS)
Description: as for outcome 3
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Strattice Reconstructive Tissue Matrix
Number analyzed (Participants) | 66
units on a scale | 83.5 (17.10)

7. Secondary Outcome: Activities Assessment Scale (AAS)
Description: as for outcome 3
Time Frame: 24 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Strattice Reconstructive Tissue Matrix
Number analyzed (Participants) | 60
units on a scale | 82.0 (17.53)

ADVERSE EVENTS:
Description: The at risk population was comprised of 80 subjects who received Strattice reinforcement of hernia repair (ITT population)
Arm/Group | Strattice
Serious Adverse Events (participants affected / at risk) | 50/80
Other Adverse Events (participants affected / at risk) | 20/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Strattice (N=80)
Abdominal Pain (Gastrointestinal disorders) | 1 (2)
Abdominal abscess (Infections and infestations) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 2 (3)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 2 (2)
Anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
Arteriosclerosis obliterans (Vascular disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Bacteraemia (Infections and infestations) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (3)
Cholecyctitis (Hepatobiliary disorders) | 2 (2)
Cholecyctitis chronic (Hepatobiliary disorders) | 1 (1)
Clostridium difficile toxin test positive (Investigations) | 1 (1)
Colostomy infection (Infections and infestations) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (5)
Delirium (Psychiatric disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Iatrogenic injury (Injury, poisoning and procedural complications) | 1 (1)
Ileus (Gastrointestinal disorders) | 5 (5)
Ileus paralytic (Gastrointestinal disorders) | 1 (1)
Incision site haematoma (Injury, poisoning and procedural complications) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 7 (7)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Metabolic disorder (Metabolism and nutrition disorders) | 1 (1)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2)
Osteomyelitis (Infections and infestations) | 1 (1)
Pancreatic fistula (Gastrointestinal disorders) | 1 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Pelvic abscess (Infections and infestations) | 2 (2)
Peripheral ischaemia (Vascular disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (3)
Post procedural fistula (Injury, poisoning and procedural complications) | 1 (1)
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Seroma (Injury, poisoning and procedural complications) | 4 (4)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (6)
Small intestinal stenosis (Gastrointestinal disorders) | 1 (1)
Suture related complication (Injury, poisoning and procedural complications) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (1)
Wound abscess (Infections and infestations) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Wound infection (Infections and infestations) | 9 (11)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Strattice (N=80)
Seroma (Injury, poisoning and procedural complications) | 20 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No